CLINICAL TRIAL: NCT04808869
Title: Effectiveness of Blood Flow Restriction During Aerobic Cycling Exercise on Balance, Knee Stability, Strength, and Aerobic Performance in Healthy Adults
Brief Title: Effectiveness of Blood Flow Restriction During Aerobic Cycling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Principal Investigator, Alexis Ortiz, Professor, University of the Incarnate Word
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0891
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Exercise Intervention
Keywords: exercise; cycle ergometer; strength
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Sham Comparator): Cycling at 70 rpm 3 times/week without any blood flow restriction cuffs
  Interventions: Other: Exercise
- BRF 60% Unilateral (Experimental): Cycling at 70 rpm 3 times/week with blood flow restriction cuffs at 60% occlusion in one leg.
  Interventions: Other: Exercise
- BFR 80% Unilateral (Experimental): Cycling at 70 rpm 3 times/week with blood flow restriction cuffs at 80% occlusion in one leg.
  Interventions: Other: Exercise
- BFR Bilateral 60% (Experimental): Cycling at 70 rpm 3 times/week with blood flow restriction cuffs at 60% occlusion in both legs.
  Interventions: Other: Exercise
- BFR 80% Bilateral (Experimental): Cycling at 70 rpm 3 times/week with blood flow restriction cuffs at 80% occlusion in both legs.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Cycling 3 times a week for 15 minutes at 70 rpm using blood flow restriction cuffs at different occlusions.
  Other Names: Blood flow restriction training

SUMMARY:
Blood flow restriction (BFR) training has become a popular alternate rehabilitation modality, intending to improve muscle strength, hypertrophy, metabolic response, and functional outcomes in diverse populations. However, there is a paucity of research evidence on the effectiveness of using BFR during aerobic exercise. Most BFR interventions have used BFR cuffs in two to four limbs, however, it is unknown if using BFR cuffs in a single limb instead of multiple limbs can produce the desired outcomes in muscle physiology and muscular adaptations. Therefore, we have divided the purpose of this study into the following three aims:

Compare physical performance measures of balance, isokinetic muscle strength, knee stability, and aerobic capacity between cycling exercise with and without BFR.

Compare physical performance measures between performing cycling exercise at 60% versus 80% blood flow occlusion.

Compare physical performance measures between bilateral BFR versus single-leg BFR during a cycling protocol.

These aims will be accomplished by randomizing 55 participants into five groups of eleven participants each: 1) control; 2) bilateral BFR cuffs with 60% occlusion; 3) bilateral BFR cuffs with 80% occlusion; 4) single-limb BFR with 60% occlusion; and 5) single-limb BFR with 80% occlusion. All participants will undergo balance, isokinetic knee strength, knee stability, and aerobic testing at baseline, 3-week, and 6-week follow-ups. The intervention for all groups will consist of 15 minutes cycling on a stationary ergometer at 70 revolutions/minute. A within- and between-group (5) by time (3) repeated measures analysis of variance (ANOVA) will be used to explore differences between group and time in addition to the interaction between these two.

DETAILED DESCRIPTION:
Experimental Design & Sample Size: This study is a randomized controlled trial with five groups of 11 participants each (N=55). Sample size was estimated with GPower using a 5-group within- and between-groups repeated measures design with three follow-up visits (0, 3, 6 weeks) yielding a power greater than 80% including 10% in attrition or missing data. Population: Healthy adults between the ages of 21-35 will be recruited. Recruitment will be as close to an equal amount of women and men as possible for all groups as the participation of women in intervention studies assessing the effectiveness of BFR training has been documented to be no more than 17%. Other criteria for participation in the study will be committing to the training and testing sessions, being in good health, and familiarization with physical activity and exercise, including riding a stationary bicycle. Participants will be excluded if they have any of the following: 1) suffered a musculoskeletal injury in the lower extremities or lower back in the past three months, 2) any contraindication to aerobic exercise testing as determined by The American College of Sports Medicine [12], 3) any contraindication to blood flow restriction training, 4) meeting or exceeding the recommended ACSM exercise guidelines of aerobic exercise 5-times/week for >20 minutes and strengthening exercise > 2-days/week [12], and 5) pregnancy for female participants (self-reported). Each participant will be required to read and sign an informed consent document approved by the Institutional Review Board before enrolling in the study and any testing being performed. The 55 participants in the five groups of 11 participants will be randomized by using a random number generator. The five groups will be randomized as follows: 1) control (Con), 2) 60% bilateral occlusion BFR (60BILAT), 3) 80% bilateral occlusion BFR (80BILAT), 60% unilateral BFR occlusion (60UNIT), and 80% unilateral BFR occlusion (80UNIT).

Instrumentation & Outcomes: Single leg balance will be measured using a Balance System SD (Biodex Medical Systems, Inc, Shirley, NY). This device measures static and dynamic multidirectional balance by the use of the validated Balance Error Scoring System (BESS) by measuring sway with eyes closed in the following conditions: 1) double-leg firm surface, 2) single-leg firm surface, 3) tandem stance firm surface, and 4) repeating the previous tests on a foam (unstable) surface. Balance and postural stability are fundamental components of athletic performance and activities of daily living making its assessment imperative to measure changes during different conditions such as injury, fatigue, concussions, etc. Furthermore, recent evidence suggests that BFR training improves balance in functional activities, but the only evidence is in the population of older adults. Knee stability will be measured during a 5-repetition single-leg step down from a 30-cm step platform with a 10-camera (120Hz sampling rate) motion analysis capture system (Qualisys AB, Göteborg, Sweden) time-synchronized to a wireless electromyography (EMG) system (Trigno, Delsys, Inc., Natick, MA). EMG data will be collected through three pre-amplified (Ag) electrodes (Trigno, Delsys Inc., Natick, MA; Bandwidth: 450 ± 50 Hz > 80 dB/dec; overall channel noise: <0.75uV) bilaterally from the vastus medialis, rectus femoris, and vastus lateralis at 2kHz and filtered through a 2nd order Butterworth filter. Knee stability is an essential outcome in rehabilitation as it is the foundation for proper alignment to prevent injuries [14], while muscle activation is one of the main constraints to knee instability, helping to prevent injuries. Given there is evidence showing BFR training increases muscle recruitment and muscular activation by the use of EMG it is imperative to determine if such improvements translate into better motor control and knee stability during functional activities. Muscle strength of the quadriceps and hamstrings will be measured with an isokinetic dynamometer (System 4 Pro, Biodex Medical Systems, Inc, Shirley, NY) at the speeds of 60˚ and 180˚ degrees per second. The dynamometer will be calibrated according to the manufacturer's recommendations. Several investigations have found improvements in isokinetic strength after BFR training. Therefore, assessment of muscle strength via isokinetic dynamometer will allow to make comparisons between the study and the current literature. Aerobic Capacity will be measured during a cycle ergometer protocol in a stationary ergometer (Velotron, Quarq Technology, Spearfish, SD) while connected to a gas analyzer (TruOne 2400, Parvomedics, Salt Lake City, UT) for the assessment of oxygen consumption [VO2 (ml/min)]. This is an exploratory outcome as aerobic exercise in a cycle exercise for 15 minutes is not expected to improve cardiovascular metabolic performance. However, Abe et al 2010 reported improvements in VO2max with a similar protocol to this study of 15 minutes of cycling with BFR cuffs. Thus, by evaluating VO2, the study will be able to determine if there is any benefit of BFR training during aerobic exercise and compare our results to the small cycling evidence with BFR cuffs.

Procedures: After consenting to participation, demographic and anthropometric information will be recorded. After measurements, participants will be equipped with retroreflective markers per Qualisys CAST model, using appropriate hypoallergenic double-side retroreflective markers for individual markers and elastic bandages with Velcro for retroreflective casts. EMG electrode placement will follow a standardized setup previously published by Ortiz et al. To minimize the effects of fatigue in task performance, the order of testing will remain constant in the following order: 1) BESS, 2) single-leg step down, 3) isokinetic testing, and 4) aerobic capacity. For the BESS, the order of the testing will be according to the protocol displayed on the platform's computer screen. Participants will perform all tests with eyes closed for 20 seconds with 10-seconds rest between conditions. Each participant will first perform the three stable conditions (double-leg, single-leg, tandem) followed by the same conditions after placing a 6cm thick foam pad over the balance platform. A special note for those participants in the single-leg BFR group will be written, denoting which leg was used for the BFR cuffs. The single-leg step-down will be performed from a 30-cm step for three 5-steps repetitions per leg, alternating legs. Each participant will stand initially on the step with both feet on the step. Upon the command "go," they will lift the corresponding leg and step down touching the floor (force plate) with the non-weight-bearing leg and will return to the original stance position. This process will be performed continuously five consecutive times. Valgus motion will be tracked with the 3-dimensional motion system and EMG through the entirety of the five single-leg stance time epochs. Valgus will be measured at the point where the participant touches the force plate. The highest valgus and EMG amplitude (RMS) of the three middle trials will be considered for analysis. A special note for those participants in the single-leg BFR group will be written, denoting which leg was used for the BFR cuffs. For the fatigue analyses, the average of the five trials for motion analysis and the entire frequency of the EMG signal will be considered for analysis. Muscle strength assessment of the quadriceps and hamstrings will follow the step-down assessment. Each participant will be seated in the dynamometer based on standardized positions. The right leg will be tested first, followed by the left one. For those participants in the single-leg BFR group, a special note will be written denoting which leg was used for the BFR cuffs. The standardized protocol set by the dynamometer computer will be followed with 60˚ and 180˚ per second. A familiarization warm-up of three to five repetitions at each speed will be performed previous to the testing at each speed, followed by a minute of rest. A total of five contractions will be performed at 60˚/second and 10 repetitions at 180˚/second. Aerobic capacity will be assessed through a standardized maximal cycle ergometer protocol. VO2 max, VO2 peak, and heart rate will be measured directly from the metabolic analyzer during this protocol. After a 10-minute rest to obtain resting heart rate, participants will start pedaling at 70 rev/min with a load of 25 Watts. Heart rate (HR) will be monitored continuously in real-time and the heart rate at the end of the first three minutes will be used to determine further load increases. The test will continue until the participant reaches one or more of the following criteria: reaches 80% of their predicted heart rate by using the heart rate reserve formula; (([220-age] -resting heart rate) x 80%) + resting heart rate, reaches an RER >1.0, or there is a leveling of the oxygen curve. Intervention: Control group: the control group will perform 15 minutes of cycling in a stationary cycle ergometer at 70 rev/min three times a week for six weeks. Subjects will wear a polar heart rate monitor through the training to record their heart rate response during the 15 minutes of training. BFR groups: all four BFR groups will perform the same training as the control group while using the BFR cuffs. This training program follows the recommendations for stationary cycling while wearing BFR cuffs of 45-60 minutes per week. Each participant in the BFR group will undergo the protocol defined by Delfi (Delfi Medical Innovations, Inc., Vancouver BC, Canada), consisting of placing the BFR cuff in the upper part of the thigh while the participant is lying supine on a table against gravity to determine full occlusion then to derived the percentage of desired occlusion (60% or 80%).

Data Analysis: Data will be screened for normality, homoscedasticity, and outliers. Independent t-tests will be performed to compared demographic (age, weight, height, BMI) variables between groups. A within- and between-group (5) by time (3) repeated measure ANOVA with interactions will be used to compare groups for all outcomes of interest. Post-hoc analyses will be used to follow up significant differences between groups, time, and the group by time interaction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 21-35.
* Committing to the training and testing sessions.
* Being in good health, and familiarization with physical activity and exercise.

Exclusion Criteria:

* Suffered a musculoskeletal injury in the lower extremities or lower back in the past three months.
* Any contraindication to aerobic exercise testing as determined by The American College of Sports Medicine.
* Any contraindication to blood flow restriction training.
* Meeting or exceeding the recommended ACSM exercise guidelines of aerobic exercise 5-times/week for >20 minutes and strengthening exercise > 2-days/week.
* Pregnancy for female participants (self-reported).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Knee valgus | 12-week
  Medial deviation of the knee during a single leg step down.
Single leg balance | 12-week
  Single leg balance on balance platform with eyes open and eyes closed for 20 seconds each.
Isokinetic strength | 12-week
  Quadriceps and hamstring strength at three different speeds; 60, 180, 300 degrees per second.
Oxygen consumption during bicycle exercise protocol | 12-week
  VO2 peak during graded cycling protocol

CONTACTS AND LOCATIONS:
Locations (1):
- School of physical Therapy-University of The Incarnate Word, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No